CLINICAL TRIAL: NCT03223285
Title: Diaphragm's Manual Therapy Reduce Pain in Patients With Chronic Neck Pain: a Randomised Controlled Trial
Brief Title: Diaphragm's Manual Therapy in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Marco Da Roit, PT, MSc, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pilota_cervicalgia_diaframma
Record Dates: First submitted 2017-07-04; First posted 2017-07-21 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Neck Pain
Keywords: Cervical spine;; Diaphragm;; Manual Therapy; Pain; Range of Motion
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Treatment Group (Experimental): Patients included in this group will receive 3 multifaced physiotherapy/osteopathic treatments + experimental manoeuvres, 1 treatment/week. Each session will last about 30 minutes.
  Interventions: Behavioral: Real Treatment Group
- Sham Treatment Group (Sham Comparator): Patients included in this group will receive 3 multifaced physiotherapy/osteopathic treatments + sham manoeuvres, 1 treatment/week. Each session will last about 30 minutes.
  Interventions: Behavioral: Sham Treatment Group

INTERVENTIONS:
Behavioral: Real Treatment Group — Real Diaphragm manoeuvres The experimental manoeuvres include the Doming The Diaphragm Technique as described by Digiovanna (2004), Chila (2011) and Yao (2014) and the Manual Diaphragm Release Technique as described by Ricard (2009), De Coster (2005) and Roha (2015). Both manoeuvres are performed in two sets of 10 repetitions, within a 1-minute interval.
  Multifaced physiotherapy/osteopathic treatment includes: vertebral mobilisations (C0-D1), high-velocity low-amplitude (HVLA) thrusts of the cervical spine, soft tissue techniques
  Arms: Real Treatment Group
Behavioral: Sham Treatment Group — Sham Diaphragm manoeuvre: the physiotherapist will simply lie hands on the rib cage, and rest along the anterolateral costal margin below rib 7, during normal breathing of the patient for 40 breathes.
  Multifaced physiotherapy/osteopathic treatment includes: vertebral mobilisations (C0-D1), high-velocity low-amplitude (HVLA) thrusts of the cervical spine, soft tissue techniques
  Arms: Sham Treatment Group

SUMMARY:
The aim of this study is to evaluate the effect of diaphragm's manual therapy in addition to cervical spine manual therapy in terms of pain, cervical spine range of motion, trigger points pain pressure threshold, disability and quality of life in patient with chronic aspecific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain since at least 3 months
* Age > 18 years and < 65 years
* Male or Female

Exclusion Criteria:

* Pregnancy
* Contraindications for manual therapy or inability to complete the treatment
* Patients who received a physiotherapy or osteopathic treatment during the last 3 months
* Medical diagnosis of rheumatologic disease
* Medical diagnosis of respiratory disease (COPD, asthma)
* Spine surgery
* Medical diagnosis of past or present cancer
* Thoracic or abdominal surgery in the last 3 years
* Whiplash injuries
* Previous cervical fracture
* Cervical anatomical changes
* Thrombotic events
* Body temperature greater than 37 degrees in the previous 48 hours
* Obesity (BMI greater than 30)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) | Week 0, 1, 2, 3, 13, 25
  The NPRS is an 11-point scale from 0-10 (0 = no pain; 10 = the most intense pain imaginable).
  Measures the subjective intensity of pain. Patients verbally select a value that is most in line with the intensity of pain that they have experienced in the last 24 hours.

SECONDARY OUTCOMES:
Change in Range of motion (ROM) | Week 0, 1, 2, 3, 13, 25
  Using the Baseline Bubble Inclinometer (Mayer 1993, Cleland, 2006), placed on the vertex of the head, taken the ROM with the patient sitting straight (flexion, extension and lateral inclinations) and supine (rotations).
Change in Pain pressure threshold | Week 0, 1, 2, 3, 13, 25
  Using a LIZARD Ahi-o-meter (CE), the change of the pain on the trigger points is measured, with the patient in sitting position, in upper trapezium and sternocleidomastoid muscle bilaterally, by the detection of trigger points from a map.
Change in Neck Disability Index (NDI) | Week 0, 3, 13, 25
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain.
Change in Medical outcomes study short form 36 (SF-36) | Week 0, 3, 13, 25
  The SF-36 is a generic patient-reported outcome measure aimed at quantifying health status, and is often used as a measure of health-related quality of life.
Adverse events | Week 2, 3, 13, 25
  Through an interview, potential adverse effects are evaluated during and after the physiotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Da Roit, PT, MSc, Principal Investigator — Università degli Studi di Ferrara, Physiotherapy Degree Course; Giulia Simoni, PT, OMT, MSc, Principal Investigator — Università degli Studi di Ferrara, Physiotherapy Degree Course
Locations (1):
- Fisiotech - Studio Associato di Fisioterapia, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simoni G, Bozzolan M, Bonnini S, Grassi A, Zucchini A, Mazzanti C, Oliva D, Caterino F, Gallo A, Da Roit M. Effectiveness of standard cervical physiotherapy plus diaphragm manual therapy on pain in patients with chronic neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:481-491. doi: 10.1016/j.jbmt.2020.12.032. Epub 2021 Feb 16. PMID 33992285